CLINICAL TRIAL: NCT04698447
Title: Effects of the Natural Supplement CitraVes Containing Nanovesicles Delivered From Citrus Limon (L.) Juice on Cardio-metabolic Risk Factors in Subjects With Metabolic Syndrome
Brief Title: The Role of a Natural Product, Containing Nanovesicles From Citrus Limon (L.) Juice, on Different CV Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Giuseppe Montalto, MD, Full Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Natural Supplement CitraVes
Record Dates: First submitted 2020-12-27; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Syndrome; Healthy Volunteers
Keywords: cardiovascular risk; extracellular vesicles; metabolic parameters; nutraceuticals; Citrus limon (L.)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Supplement blinded (Experimental): 20 subjects with the metabolic syndrome receiving natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice (1000 mg/day)
  Interventions: Dietary Supplement: Natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice_MetS
- Placebo blinded (Placebo Comparator): 20 subjects with the metabolic syndrome receiving placebo (without any active ingredients)
  Interventions: Dietary Supplement: Placebo (without any active ingredients)
- Dietary Supplement open-label (Active Comparator): 20 healthy volunteers receiving natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice (1000 mg/day)
  Interventions: Dietary Supplement: Natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice_HS

INTERVENTIONS:
Dietary Supplement: Natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice_MetS — 20 eligible subjects with the metabolic syndrome (MetS) will take natural supplement containing a spray-dried formulation of citraVes™, directly in the mouth, without water, to be dissolved preferably under the tongue, at a stable dose of one sachet a day (1000 mg/day) for 6 months and as add-on therapy to the ongoing treatment, maintained at fixed doses for the entire study.
  Arms: Dietary Supplement blinded
Dietary Supplement: Placebo (without any active ingredients) — 20 eligible subjects with the metabolic syndrome will take placebo in a spray-dried formulation (without any active ingredients) directly in the mouth, without water, to be dissolved preferably under the tongue, at a stable dose of one sachet a day for 6 months, as add-on therapy to the ongoing treatment, maintained at fixed doses for the entire study.
  Arms: Placebo blinded
Dietary Supplement: Natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice_HS — 20 eligible healthy subjects (HS) will take natural supplement containing a spray-dried formulation of citraVes™, directly in the mouth, without water, to be dissolved preferably under the tongue, at a stable dose of one sachet a day (1000 mg/day) for 6 months, maintained at fixed doses for the entire study.
  Arms: Dietary Supplement open-label

SUMMARY:
Clinical trial about beneficial effects of natural supplement in a spray-dried formulation, citraVes™, obtained from Citrus Limon (L.) juice on general body health.

DETAILED DESCRIPTION:
This is one randomized, double-blind, placebo-controlled study. The aim of the present study is to investigate the role of a natural product, citraVes™ on several cardiovascular risk factors.

The research hypothesis is to evaluate whether this natural supplement containing nanovesicles delivered from Citrus Limon (L.) juice (Navhetec S.R.L., Palermo, Italy) may improve different cardio-metabolic parameters in subjects with the metabolic syndrome. All subjects will be evaluated at baseline, after 1 month and after 3 and 6 months of supplementation with natural product or placebo.

ELIGIBILITY:
Inclusion Criteria:

* men and women > 18 years old;
* body mass index (BMI) > 25 kg/m²;
* subjects who are able to swallow;
* subjects who are willing to participate in the study and therefore, to sign informed consent prior to any study procedure;
* the inclusion criteria for patients with MetS was also the diagnosis of MetS, as defined by international consensus [Alberti KG, et al. Circulation. 2009; 120:1640-5].

Exclusion Criteria:

* pregnancy or the willingness to become pregnant;
* severe renal or hepatic impairment;
* known severe infections (such as HIV, HBV, HCV)
* any neoplasms;
* the exclusion criteria for healthy volunteers were also diagnosis of any one of the following diseases: hypertension, diabetes mellitus, dyslipidaemia or metabolic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Plasma Lipids in Healthy Subjects | 3 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on low-density lipoprotein cholesterol (LDL-C), total cholesterol, triglycerides, and high-density lipoprotein cholesterol (HDL-C) (mmol/l).
Change from Baseline in Plasma Lipids in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on low-density lipoprotein cholesterol (LDL-C), total cholesterol, triglycerides, and high-density lipoprotein cholesterol (HDL-C) (mmol/l).

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference in Healthy Subjects | 3 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on waist circumference (cm).
Change from Baseline in Waist Circumference in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on waist circumference (cm).
Change from Baseline in Body Mass Index (BMI) in Healthy Subjects | 3 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on body weight (kg) and height (m) that will be combined to report BMI in kg/m^2.
Change from Baseline in Body Mass Index (BMI) in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on body weight (kg) and height (m) that will be combined to report BMI in kg/m^2.
Change from Baseline in Glycemia in Healthy Subjects | 3 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on plasma glycemia (mmol/l).
Change from Baseline in Glycemia in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on plasma glycemia (mmol/l).
Change from Baseline in Glycated Haemoglobin in Healthy Subjects | 3 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on glycated haemoglobin (HbA1c) (%).
Change from Baseline in Glycated Haemoglobin in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on glycated haemoglobin (HbA1c) (%).
Change from Baseline in Subclinical Atherosclerosis in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on subclinical atherosclerosis assessed by carotid intima-media thickness (CIMT) (mm).
Change from Baseline in Plasma Cytokines in Subjects with Metabolic Syndrome | 6 months
  Effect of natural supplement containing nanovesicles from Citrus Limon (L.) juice on plasma cytokines (inflammatory markers) (pg/ml), that will be assessed using available enzyme-linked immunosorbent assay (ELISA) kits.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Montalto, MD, Principal Investigator — University Hospital of Palermo, Palermo, Italy
Locations (1):
- University Hospital of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Abundis E, Mendez-Del Villar M, Perez-Rubio KG, Zuniga LY, Cortez-Navarrete M, Ramirez-Rodriguez A, Gonzalez-Ortiz M. Novel nutraceutic therapies for the treatment of metabolic syndrome. World J Diabetes. 2016 Apr 10;7(7):142-52. doi: 10.4239/wjd.v7.i7.142. PMID 27076875
- [Background] Corrado C, Raimondo S, Chiesi A, Ciccia F, De Leo G, Alessandro R. Exosomes as intercellular signaling organelles involved in health and disease: basic science and clinical applications. Int J Mol Sci. 2013 Mar 6;14(3):5338-66. doi: 10.3390/ijms14035338. PMID 23466882
- [Background] Lakkaraju A, Rodriguez-Boulan E. Itinerant exosomes: emerging roles in cell and tissue polarity. Trends Cell Biol. 2008 May;18(5):199-209. doi: 10.1016/j.tcb.2008.03.002. Epub 2008 Apr 7. PMID 18396047
- [Background] Wang B, Zhuang X, Deng ZB, Jiang H, Mu J, Wang Q, Xiang X, Guo H, Zhang L, Dryden G, Yan J, Miller D, Zhang HG. Targeted drug delivery to intestinal macrophages by bioactive nanovesicles released from grapefruit. Mol Ther. 2014 Mar;22(3):522-534. doi: 10.1038/mt.2013.190. Epub 2013 Aug 13. PMID 23939022
- [Background] Ju S, Mu J, Dokland T, Zhuang X, Wang Q, Jiang H, Xiang X, Deng ZB, Wang B, Zhang L, Roth M, Welti R, Mobley J, Jun Y, Miller D, Zhang HG. Grape exosome-like nanoparticles induce intestinal stem cells and protect mice from DSS-induced colitis. Mol Ther. 2013 Jul;21(7):1345-57. doi: 10.1038/mt.2013.64. Epub 2013 Jun 11. PMID 23752315
- [Background] Raimondo S, Naselli F, Fontana S, Monteleone F, Lo Dico A, Saieva L, Zito G, Flugy A, Manno M, Di Bella MA, De Leo G, Alessandro R. Citrus limon-derived nanovesicles inhibit cancer cell proliferation and suppress CML xenograft growth by inducing TRAIL-mediated cell death. Oncotarget. 2015 Aug 14;6(23):19514-27. doi: 10.18632/oncotarget.4004. PMID 26098775
- [Background] Li C, Schluesener H. Health-promoting effects of the citrus flavanone hesperidin. Crit Rev Food Sci Nutr. 2017 Feb 11;57(3):613-631. doi: 10.1080/10408398.2014.906382. PMID 25675136